CLINICAL TRIAL: NCT00186927
Title: A Phase I Study of Unmodified Live Intranasal Sendai Virus Vaccine in Children and Toddlers: Assessment of Safety and Immunogenicity
Brief Title: A Study to Assess the Safety of Live Intranasal Sendai Virus Vaccine in Children and Toddlers
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: voluntary Hold because of COVID-19, all participants were off study prior to the hold.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SENDAI
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Parainfluenza; Respiratory Viral Infections
Keywords: Vaccine; Sendai virus vaccine
MeSH Terms: conditions — Paramyxoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants will be studied in three cohorts:
  * Healthy seropositive children 3 years up to 6 years
  * Healthy seropositive toddlers 12 months up to 24 months
  * Healthy seronegative toddlers 12 months up to 24 months.
  Each cohort will receive Sendai virus vaccine.
  Interventions: Biological: Sendai virus vaccine

INTERVENTIONS:
Biological: Sendai virus vaccine — Enders strain; a live, unmodified intranasally administered Sendai virus vaccine; given once in a dose escalation study, 5 x 10^5 to 5 x 10^7 EID(50) units.

SUMMARY:
Croup is an illness of young children that is caused by a virus. With this illness, the child has fever, cough, and hoarseness. Although the illness usually gets better in 2 to 4 days, some children may be admitted to the hospital and a few infants may require an intervention to help their breathing. This illness is most often caused by a virus called parainfluenza virus type 1, but it can be caused by other viruses. The experimental vaccine that is being investigated in this study is intended to try to prevent croup caused by parainfluenza virus type 1. Currently, there are no vaccines to prevent this virus, or medications available to treat the illness once infection has occurred.

This research study is testing a new experimental live-virus vaccine that is given by placing liquid drops in the nose. The Sendai virus is very similar to the virus that causes croup, but it has never been found to cause illness in people. Previous studies in animals have shown that the vaccine provided protection against the croup virus, and did not cause illness. Many people have been exposed to the Sendai virus, but no one has been known to develop illness. Several healthy adults have been given the Sendai virus vaccine being studied, and they did not experience any serious side effects or illness.

DETAILED DESCRIPTION:
The main aim of the study is to assess the tolerance and safety of escalating doses of intranasal Sendai virus in children and toddlers.

The secondary objective of the study is to assess the magnitude and duration of the immune response elicited by intranasal Sendai virus. Responses between seropositive and seronegative children will be compared.

This study also tests the safety and immunogenicity of a booster vaccination at the highest dose tolerated during primary immunization dose-escalation.

ELIGIBILITY:
Inclusion Criteria;

* Parent or legal guardian willing and able to give informed consent and comply with study requirements
* Child is greater than or equal to one year of age and less than six years of age
* Adequate blood, liver and kidney function
* Has not or will not receive other vaccinations within 30 days of receiving study vaccine

Exclusion Criteria:

* History of allergy to eggs or gentamicin
* History of lung disease, asthma, and hospitalization for respiratory illness, immunodeficiency, sickle cell disease, or any other serious underlying condition
* Children who have a family history of primary immunodeficiency or lack history of maternal or paternal immune status
* Height or weight less than 5th percentile
* Upper respiratory tract infection (URI) or household member with URI
* Evidence of developmental delay or evolving neurological disorders
* Household member or daycare contact (i.e. stay in the same room in daycare) less than 24 months of age if same room contact is expected within 14 days of vaccination or 7 days after booster, or prior to evidence of vaccine clearance
* Immunodeficient household members or other close contacts if same room contact is expected within 14 days of vaccination or 7 days after booster, or prior to evidence of vaccine clearance
* Current use of investigational or immunosuppressive drugs (e.g., steroids)
* Current use of antibiotics or antivirals

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2005-05-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To determine if giving live Sendai virus (in the form of a vaccine) to children through their nose is safe (causes no serious illness) | 6 months after enrollment complete
To determine if a child's body responds to the presence of the Sendai virus by making proteins in the blood called antibodies that can find and kill the croup virus | 6 months after enrollment complete

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Adderson, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Adderson E, Allison KJ, Branum K, Sealy RE, Jones BG, Surman SL, Penkert RR, Hayden RT, Russell CJ, Portner A, Slobod KS, Hurwitz JL. Intranasal Sendai Virus Vaccination of Seropositive Children 1 to 2 Years of Age in a Phase I Clinical Trial Boosts Immune Responses Toward Human Parainfluenza Virus Type 1. Vaccines (Basel). 2025 Apr 19;13(4):430. doi: 10.3390/vaccines13040430. PMID 40333329
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Croup Study Volunteer Recruitment Information — https://www.stjude.org/research/clinical-trials/sendai-infectious-disease/croup-study.html
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols